CLINICAL TRIAL: NCT01763164
Title: The NEMO Trial (NRAS Melanoma and MEK Inhibitor):A Randomized Phase III, Open Label, Multicenter, Two-arm Study Comparing the Efficacy of MEK162 Versus Dacarbazine in Patients With Advanced Unresectable or Metastatic NRAS Mutation-positive Melanoma
Brief Title: Study Comparing the Efficacy of MEK162 Versus Dacarbazine in Unresectable or Metastatic NRAS Mutation-positive Melanoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMEK162A2301; C4211002 (Other: Alias Study Number); 2012-003593-51 (EudraCT Number)
Record Dates: First submitted 2013-01-04; First posted 2013-01-08 (Estimated); Results first posted 2021-03-22 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Metastatic or Unresectable Cutaneous Melanoma
Keywords: Melanoma; Cutaneous melanoma; Skin disease; Skin cancer; Skin Neoplasms; Neoplasm Metastasis
MeSH Terms: conditions — Neoplasm Metastasis; Melanoma; Skin Diseases; Skin Neoplasms | interventions — binimetinib; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MEK162 (Experimental)
  Interventions: Drug: MEK162
- Dacarbazine (Active Comparator)
  Interventions: Drug: Dacarbazine

INTERVENTIONS:
Drug: MEK162 — MEK162 will be administered as a fixed dose of 45 mg (3 x 15 mg tablets) BID, with a glass of water and taken with or without food.
  Arms: MEK162
Drug: Dacarbazine — Patients randomized to dacarbazine will receive an IV infusion of dacarbazine 1000 mg/m2 over the course of 1 hour on day 1 and then every three weeks.
  Arms: Dacarbazine

SUMMARY:
Two-arm, randomized, prospective, open-label, multi-center, phase III study to compare the efficacy and safety of MEK162 (45 mg BID) versus dacarbazine (1000 mg/m2 IV every 3 weeks) in patients with advanced (Stage IIIC) unresectable or metastatic (Stage IV) NRAS Q61 mutation-positive cutaneous or unknown primary melanoma. The mutation analysis will be performed at a central laboratory. Only those patients with Q61 mutation per central laboratory and meet all eligibility criteria will be randomized. A total of 393 patients will be randomized 2:1 to receive either MEK162 or dacarbazine. Patients will be stratified according to AJCC stage (IIIC, IVM1a, and IVM1b versus IVM1c), ECOG Performance status (0 versus 1) and any prior number of lines of immunotherapy (immunotherapies versus none). This study will use an Interactive Response Technology (IRT). The primary end point of the study is progression-free survival. Key secondary end point is overall survival

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of locally advanced, unresectable or metastatic cutaneous or melanoma of unknown primary AJCC Stage IIIC or IV (uveal and mucosal melanoma are excluded)
* Presence of NRAS Q61 mutation in tumor tissue prior to randomization as determined by a Novartis designated central laboratory
* Naïve untreated patients or patients who have progressed on or after any number of prior lines of immunotherapy for unresectable locally advanced or metastatic melanoma
* Evidence of at least one measurable lesion as detected by radiological or photographic methods
* Adequate bone marrow, organ function, cardiac and laboratory parameters
* Normal functioning of daily living activities

Exclusion Criteria:

* Any untreated CNS metastases
* Uveal or mucosal melanoma
* History of or current evidence of retinal vein occlusion (RVO) or risk factors of RVO
* Patients with washout period < 6 weeks from the last dose of ipilimumab or other immunotherapy.
* Previous systemic chemotherapy for unresectable locally advanced or metastatic melanoma.
* History of Gilbert's syndrome
* Prior therapy with a MEK- inhibitor
* Impaired cardiovascular function or clinically significant cardiovascular diseases
* Uncontrolled arterial hypertension despite medical treatment
* HIV positive or active Hepatitis A or B
* Impairment of gastrointestinal function
* Patients who have undergone major surgery or radiotherapy ≤ 3 weeks prior to starting study drug or who have not recovered from side effects of such procedure;
* Patients with neuromuscular disorders that are associated with elevated CK.
* Pregnant or nursing (lactating) women
* Medical, psychiatric, cognitive or other conditions that may compromise the patient's ability to understand the patient information, give informed consent, comply with the study protocol or complete the study

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2013-07-12 (Actual); Primary Completion 2015-12-01 (Actual); Study Completion 2019-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (220):
- United States (69):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Highlands Oncology Group, Rogers, Arkansas
  - Florida Cancer Specialists, Altamonte Springs, Florida
  - Florida Cancer Specialists, Bonita Springs, Florida
  - Florida Cancer Specialists, Bradenton, Florida
  - Florida Cancer Specialists, Brandon, Florida
  - Florida Cancer Specialists, Cape Coral, Florida
  - Florida Cancer Specialists, Clearwater, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Cancer Specialists, Gainesville, Florida
  - Florida Cancer Specialists, Hudson, Florida
  - Florida Cancer Specialists, Inverness, Florida
  - Florida Cancer Specialists, Largo, Florida
  - Florida Cancer Specialists, Naples, Florida
  - Florida Cancer Specialists, New Port Richey, Florida
  - Florida Cancer Specialists, Orange City, Florida
  - Florida Cancer Specialists, Orlando, Florida
  - Florida Cancer Specialists, Port Charlotte, Florida
  - Florida Cancer Specialists, Sarasota, Florida
  - Florida Cancer Specialists, Spring Hill, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Florida Cancer Specialists, Tampa, Florida
  - Florida Cancer Specialists, Tavares, Florida
  - Florida Cancer Specialists, Venice, Florida
  - Oncology Specialists, SC, Niles, Illinois
  - Oncology Specialists, SC, Park Ridge, Illinois
  - Goshen Center For Cancer Care, Goshen, Indiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Harry and Jeannette Weinberg Cancer Institute @Franklin Square, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Kresge Eye Institute, Bingham Farms, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Kresge Eye Institute, Detroit, Michigan
  - Karmanos Cancer Institute of Farmington Hills, Farmington Hills, Michigan
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Cooper University Hospital, Voorhees Township, New Jersey
  - The Ohio State University James Cancer Hospital, Columbus, Ohio
  - The Ohio State University Martha Morehouse Medical Plaza, Columbus, Ohio
  - OHSU Knight Cancer Institute, Portland, Oregon
  - Kaiser Permanente Northwest Region Oncology/Hematology, Portland, Oregon
  - OHSU Center for Health and Healing, Portland, Oregon
  - OHSU, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Cancer Center Associates - Medical Oncology, Allentown, Pennsylvania
  - St. Luke's Cancer Center - Allentown Campus, Allentown, Pennsylvania
  - St. Luke's Hospital - Allentown Campus, Allentown, Pennsylvania
  - Cancer Center Associates - Medical Oncology, Bethlehem, Pennsylvania
  - St. Luke's University Hospital - Bethlehem Campus, Bethlehem, Pennsylvania
  - St. Luke's Cancer Center - Anderson Campus, Easton, Pennsylvania
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania, Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Thomas Jefferson Medical Oncology, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - St. Luke's Hospital - Quakertown Campus, Quakertown, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology-Austin Central, Austin, Texas
  - Elliot J. Ginchansky, MD, PA, Dallas, Texas
  - Dennis B. Kay, Dallas, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern University Hospital- St. Paul, Dallas, Texas
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - UT Southwestern Medical Center at Dallas, Dallas, Texas
  - UT Southwestern University Hospital - Zale Lipshy, Dallas, Texas
  - US Oncology, Fort Worth, Texas
  - US Oncology, The Woodlands, Texas
- Argentina (4):
  - Sanatorio de La Providencia, Buenos Aires, Ciudad Autónoma de Buenosaires
  - Centro de Investigación Clínica ? Clínica Viedma, Viedma, Río Negro Province
  - Centro Oncologico de Rosario, Rosario, Santa Fe Province
  - Fundacion CIDEA, Buenos Aires
- Australia (5):
  - Chris O'Brien Lifehouse Hospital, Camperdown, New South Wales
  - Lake Macquarie Private Hospital, Gateshead, New South Wales
  - Melanoma Institute Australia, North Sydney, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
- Austria (4):
  - LKH-Universitätsklinikum Klinikum Graz, Graz, Styria
  - Universitätsklinikum Innsbruck, Innsbruck, Tyrol
  - Salzburger Landeskliniken, Salzburg
  - Allgemeines Krankenhaus der Stadt Wien, Vienna
- Belgium (3):
  - Sint-Augustinuskliniek, Wilrijk, Antwerpen
  - UZ Gasthuisberg, Leuven
  - CHU Sart Tilman, Liège
- Brazil (4):
  - Hospital de Clinicas de Passo Fundo, Passo Fundo, Rio Grande do Sul
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - INCA Instituto Nacional de Cancer, Rio de Janeiro
  - Hospital São José, São Paulo
- Canada (6):
  - Alberta Health Services - Cross Cancer Institute, Edmonton, Alberta
  - London Regional Cancer Program, London, Ontario
  - Sunnybrook Research Institute Centre, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - McGill University Health Center / Royal Victoria Hospital, Montreal, Quebec
  - CHU de Quebec - L'Hotel-Dieu de Quebec, Québec
- Czechia (4):
  - Mou/Mmci - Ppds, Brno, South Moravian
  - Fakultni nemocnice Ostrava, Ostrava
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Vseobecna Fakultni Nemocnice V Praze, Prague
- France (12):
  - CHU Angers, Angers, Maine-et-loire
  - CHRU de Lille - Hôpital Huriet, Lille, NORD
  - Centre Léon Bérard Centre Régional de Lutte Contre Le Cancer Rhône Alpes, Lyon, Rhône
  - Hôpital Saint-André, Bordeaux
  - Centre Hospitalier Universitaire Ambroise Pare, Boulogne-Billancourt
  - Centre Hospitalier Le Mans, Le Mans
  - Hopitaux de La Timone, Marseille
  - Groupe Hospitalier Archet I Et II, Nice
  - Hôpital Saint Louis, Paris
  - Service de PneumologieCHU Lyon Sud, Pierre-Bénite
  - Hôpital Robert Debré, Reims
  - Centre Hospitalier Universitaire Hopitaux de Rouen, Rouen
- Germany (25):
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Klinikum Mannheim Universitätsklinikum gGmbH, Mannheim, Baden-Wurttemberg
  - LMU Klinikum der Universität München, München, Bavaria
  - University Clinic Regensburg - PPDS, Regensburg, Bavaria
  - Universitätsklinikum Würzburg, Würzburg, Bavaria
  - Institut für Diagnostische und Interventionelle Radiologie Frankfurt, Frankfurt am Main, Hesse
  - Universitätsklinikum Frankfurt, Frankfurt am Main, Hesse
  - Elben Klinken Stade Buxtehude, Buxtehude, Lower Saxony
  - Johannes Wesling Klinikum Minden, Minden, North Rhine-Westphalia
  - Universitatsklinikum Leipzig, Leipzig, Saxony
  - Klinikum Dorothea Christiane Erxleben Quedlinburg GmbH, Quedlinburg, Saxony-Anhalt
  - Charite Campus Mitte, Berlin, Schleswig-Holstein
  - Helios Klinikum Erfurt, Erfurt, Thuringia
  - Uniklinik Köln, Cologne
  - Universitätsklinikum Carl Gustav Carus an der TU Dresden, Dresden
  - Universitätsklinikum Essen, Essen
  - SRH Wald-Klinikum Gera GmbH, Gera
  - Medizinische Hochschule Hannover (Hannover Medical School), Hanover
  - University Clinic Heidelberg - PPDS, Heidelberg
  - Universitatsklinikum Schleswig-Holstein, Kiel
  - Universitatsklinikum Schleswig-Holstein, Lübeck
  - Fachklinik Hornheide, Münster
  - Klinikum Nuernberg Nord, Nuremberg
  - Universitätsklinikum Tübingen, Tübingen
  - Universit*ätsklinikum Ulm, Ulm
- Laiko General Hospital of Athens, Athens, Greece
- Hungary (4):
  - Magyar Honvédség Egészségügyi Központ, Budapest
  - Orszagos Onkologiai Intezet, Budapest
  - Somogy Megyei Kaposi Mór Oktató Kórház, Kaposvár
  - Jasz-Nagykun-Szolnok Megyei Hetenyi Geza Korhaz-Rendelointezet, Szolnok
- Israel (3):
  - Rambam Medical Center - PPDS, Haifa
  - Hadassah Medical Center - PPDS, Jerusalem
  - Sheba Medical Center - PPDS, Ramat Gan
- Italy (13):
  - AOU dell'Università degli Studi della Campania Luigi Vanvitelli, Napoli, Campania
  - Istituto Dermopatico dell'Immacolata IRCCS, Rome, Lazio
  - ASST degli Spedali Civili di Brescia - Spedali Civili di Brescia, Brescia, Lombardy
  - Istituto Nazionale per lo studio e la cura dei tumori Fondazione Giovanni Pascale, Napoli, Naples
  - Istituto Oncologico Veneto - I.R.C.C.S., Padua, Veneto
  - IRCCS Giovanni Paolo II Istituto Oncologico, Bari
  - ASST Papa Giovanni XXIII - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - IRCCS Az. Osp. Universitaria San Martino- IST, Genova
  - Ospedale San Raffaele S.r.l. - PPDS, Milan
  - Fondazione IRCCS 'Istituto Nazionale dei Tumori' di Milano, Milan
  - Istituto Nazionale Tumori Regina Elena, Roma
  - Azienza Ospedaliera Universitaria Senese, Siena
  - A.O.U. Città della Salute e della Scienza di Torino - Presidio S. Lazzaro, Torino
- Japan (3):
  - Shinshu University Hospital, Matsumoto, Nagano
  - National Cancer Center Hospital, Chūōku
  - Kansai Medical University Hospital, Hirakata
- Netherlands (4):
  - Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland
  - Het Nederlands Kanker Instituut Antoni Van Leeuwenhoek Ziekenhuis, Amsterdam, North Holland
  - Leids Universitair Medisch Centrum, Leiden, South Holland
  - Isala Klinieken, Zwolle
- Poland (3):
  - Centrum Medyczne MAVIT Sp. z o.o., Warsaw, Masovian Voivodeship
  - Lux Med, Warsaw
  - Centrum Onkologii Instytut im. Marii Sklodowskiej-Curie, Warsaw
- Portugal (4):
  - Instituto Português de Oncologia de Lisboa Francisco Gentil, E.P.E., Lisbon, Lisbon District
  - Hospital Garcia de Orta*E.P.E., Almada
  - Centro Hospitalar Lisboa Norte, E.P.E. - Hospital de Santa Maria, Lisbon
  - Instituto Portugues de Oncologia Do Porto Francisco Gentil Epe - PPDS, Porto
- Russia (3):
  - Russian Oncology Research Center n a N N Blokhin, Moscow
  - Ryazan Regional Clinical Oncology Dispensary, Ryazan
  - Scientific Research Institute of Oncology n.a. N.N. Petrov, Saint Petersburg
- Narodny onkologicky ustav, Bratislava, Slovakia
- South Africa (5):
  - University of The Free State, Bloemfontein, Free State
  - Sandton Oncology Medical Group, Johannesburg, Gauteng
  - Sandton Oncology Medical Research, Johannesburg, Gauteng
  - Steve Biko Academic Hospital, Pretoria, Gauteng
  - Mary Potter Oncology Centre, Pretoria, Gauteng
- South Korea (4):
  - Asan Medical Center - PPDS, Seoul
  - Samsung Medical Center - PPDS, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System - PPDS, Seoul
- Spain (16):
  - ICO l'Hospitalet - Hospital Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital Regional Universitario de Malaga Hospital General, Málaga, Málaga
  - Clinica Universidad Navarra, Pamplona, Navarre
  - Hospital Universitario A Coruña, A Coruña
  - Hospital Universitario Vall d'Hebrón - PPDS, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - ICO l'Hospitalet - Hospital Duran i Reynals, Barcelona
  - Complejo Hospitalario Universitario Insular - Materno Infantil, Gran Canaria
  - Hospital General Universitario Gregorio Maranon, Madrid
  - MD Anderson Cancer Center, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario HM Sanchinarro - CIOCC, Madrid
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Virgen de La Salud, Toledo
  - Fundacion Instituto Valenciano de Oncologia, Valencia
  - Consorcio Hospital General Universitario de Valencia, Valencia
- Sweden (2):
  - Skanes Universitetssjukhus Lund, Lund, Skåne County
  - Skanes Universitetssjukhus Lund, Lund
- Switzerland (3):
  - Universitätsspital Zürich, Zurich, Zürich (DE)
  - Hôpitaux Universitaires de Genève, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
- Turkey (Türkiye) (5):
  - Ege University Medical Faculty, Bornova, İzmir
  - Adana Ba?kent Hastanesi K??la Yerle?kesi, Adana
  - Hacettepe University Medical Faculty, Ankara
  - Baskent University Medical Faculty Ankara Hospital, Ankara
  - Istanbul University Cerrahpasa Medical Faculty Hospital, Istanbul
- United Kingdom (10):
  - Bristol Haematology and Oncology Centre, Bristol, Bristol, CITY of
  - Royal Cornwall Hospital, Truro, Cornwall
  - The Royal Sussex County Hospital, Brighton, EAST Sussex
  - Broomfield Hospital, Chelmsford, Essex
  - Singleton Hospital - PPDS, Swansea, Glamorgan
  - Royal Preston Hospital, Preston, Lancashire
  - Royal Marsden Hospital - Surrey, London, London, CITY of
  - Queen Elizabeth Hospital, Birmingham
  - St James s Institute of Clinical Oncology, Leeds
  - Clatterbridge Hospital, Metropolitan Borough of Wirral

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Dummer R, Schadendorf D, Ascierto PA, Arance A, Dutriaux C, Di Giacomo AM, Rutkowski P, Del Vecchio M, Gutzmer R, Mandala M, Thomas L, Demidov L, Garbe C, Hogg D, Liszkay G, Queirolo P, Wasserman E, Ford J, Weill M, Sirulnik LA, Jehl V, Bozon V, Long GV, Flaherty K. Binimetinib versus dacarbazine in patients with advanced NRAS-mutant melanoma (NEMO): a multicentre, open-label, randomised, phase 3 trial. Lancet Oncol. 2017 Apr;18(4):435-445. doi: 10.1016/S1470-2045(17)30180-8. Epub 2017 Mar 9. PMID 28284557

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants randomized were with previously untreated, advanced unresectable or metastatic Neuroblastoma RAS viral oncogene homolog (NRAS) mutation-positive melanoma as confirmed by central assessment.
Groups:
- Binimetinib (MEK162): Participants received oral binimetinib 45 milligram (mg) (3*15 mg tablets) twice daily, until disease progression (PD), unacceptable toxicity, death, physician decision, study termination or discontinuation due to any other reason (e.g., withdrawal of consent, lost to follow-up, start of a new anti-cancer therapy). Maximum duration of binimetinib treatment exposure in the study was 215.4 weeks and participants were followed up to 30 days after last dose of study treatment. Participants who discontinued study treatment due to start of a new anti-cancer therapy, were followed up at every 9 weeks until documented progression per Blinded Independent Review Committee (BIRC), withdrawal of consent, lost to follow-up, study closure or death whichever occurred first.
- Dacarbazine: Participants received intravenous (IV) dacarbazine 1000 mg per square meter (mg/m^2) once every 3 weeks until PD, unacceptable toxicity, death, physician decision, study termination or discontinuation due to any other reason (e.g., withdrawal of consent, lost to follow-up, start of a new anti-cancer therapy). Maximum duration of dacarbazine treatment exposure in the study was 119.9 weeks and participants were followed up to 30 days after last dose of study treatment. Participants who discontinued study treatment due to start of a new anti-cancer therapy, were followed up at every 9 weeks until documented progression per BIRC, withdrawal of consent, lost to follow-up, study closure or death whichever occurred first.
Period: Treatment Phase
Arm/Group | Binimetinib (MEK162) | Dacarbazine
Started | 269 | 133
Treated/Safety Set | 269 | 114
Full Analysis Set | 269 | 133
Completed | 0 | 0
Not Completed | 269 | 133
Not completed — Participant/Guardian decision | 26 | 14
Not completed — Protocol Violation | 1 | 1
Not completed — Progressive Disease | 142 | 76
Not completed — Physician Decision | 24 | 13
Not completed — Death | 10 | 1
Not completed — Adverse Event | 66 | 8
Not completed — Randomized but not Treated | 0 | 19
Not completed — Other | 0 | 1
Period: Follow up Phase
Arm/Group | Binimetinib (MEK162) | Dacarbazine
Started | 200 (Participants were followed up after completion or discontinuation of treatment.) | 78 (Participants were followed up after completion or discontinuation of treatment.)
Completed | 3 | 3
Not Completed | 197 | 75
Not completed — New therapy for study indication | 12 | 3
Not completed — Death | 21 | 4
Not completed — Subject/guardian decision | 9 | 2
Not completed — Progressive disease | 127 | 62
Not completed — Physician Decision | 10 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Adverse Event | 17 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Binimetinib (MEK162) | Dacarbazine | Total
Number analyzed (Participants) | 269 | 133 | 402
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (12.28) | 60.6 (13.35) | 62.6 (12.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 48 | 151
  Male | 166 | 85 | 251

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Description: PFS: time from randomization to first documented PD or death due to any cause, whichever occurred first. RECIST 1.1, PD: >=20% increase in sum of diameter of target lesions (TLs) taking as reference the smallest sum on study (including baseline sum), sum must also be an absolute increase of >=5 mm; unequivocal progression of existing non-TLs; appearance of >=1 lesion. Complete response (CR): disappearance of all lesions; any pathological lymph nodes (TLs) or non-pathological (non-TLs) must have reduction in short axis to <10 mm; normalization of tumor marker level for non-TLs. Partial response (PR): >=30% decrease in sum of diameter of all TLs, referring baseline sum of diameters. Stable disease (SD): neither sufficient shrinkage to qualify for PR nor increase in lesions qualified for PD referring smallest sum diameter. With no event at time of analysis cut-off or at start of any new anti-neoplastic therapy, PFS censored at date of last adequate tumor assessment of CR, PR or SD.
Time Frame: From the date of randomization to the date of the first documented PD or death, whichever occurred first (maximum up to 77 weeks for binimetinib arm; maximum up to 61 weeks for dacarbazine arm)
Population: FAS consisted of all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Binimetinib (MEK162) | Dacarbazine
Number analyzed (Participants) | 269 | 133
Months | 2.83 [2.76 to 3.55] | 1.51 [1.48 to 1.71]
Statistical Analysis 1: Comparison: Binimetinib (MEK162) vs Dacarbazine; Hazard ratio was obtained from the stratified unadjusted Cox model. P-value was obtained from the one-sided stratified log-rank test; Test type: Superiority; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.62, 95% CI 2-sided [0.47 to 0.80]

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time from the date of randomization to the date of death due to any cause. If a participant was not known to have died, overall survival was censored at the date of last known date participant alive.
Time Frame: From the date of randomization to the date of death (maximum up to 107 weeks for binimetinib arm; maximum up to 88 weeks for dacarbazine arm)
Population: FAS consisted of all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Binimetinib (MEK162) | Dacarbazine
Number analyzed (Participants) | 269 | 133
Months | 10.97 [8.94 to 13.60] | 10.09 [7.03 to 16.46]
Statistical Analysis 1: Comparison: Binimetinib (MEK162) vs Dacarbazine; Hazard ratio was obtained from the stratified unadjusted Cox model. P-value was obtained from the one-sided stratified log rank test; Test type: Superiority; p = 0.499, Log Rank; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.75 to 1.33]

3. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR: percentage of participants with best overall response (BOR) of CR or PR. BOR: best response recorded from start of treatment until CR or PR. RECIST V1.1, a) CR: disappearance of all lesions; any pathological lymph nodes (TLs) or non-pathological (non-TLs) must have reduction in short axis to <10 mm; normalization of tumor marker level for non-TLs; b) PR: >=30% decrease in sum of diameter of all TLs, taking as reference baseline sum of diameters. ORR is reported for confirmed and unconfirmed responses. Confirmed CR or PR = at least 2 determinations of CR or PR at least 4 weeks apart before PD. PD: >=20% increase in sum of diameter of all measured target lesions, taking as reference smallest sum of diameter of all TLs recorded at or after baseline, sum must also be absolute increase of >=5 mm. Unequivocal progression of existing non TLs. Appearance of at least 1 new lesion.
Time Frame: From date of randomization until first documented response of CR or PR (maximum up to 77 weeks for binimetinib arm; maximum up to 61 weeks for dacarbazine arm)
Population: FAS consisted of all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Binimetinib (MEK162) | Dacarbazine
Number analyzed (Participants) | 269 | 133
Percentage of Participants
  Confirmed ORR | 15.2 [11.2 to 20.1] | 6.8 [3.1 to 12.5]
  Confirmed + Unconfirmed: ORR | 22.7 [17.8 to 28.2] | 9.8 [5.3 to 16.1]
Statistical Analysis 1: Comparison: Binimetinib (MEK162) vs Dacarbazine; Confirmed ORR: The p-value (2-sided) was computed from stratified Cochran-Mantel-Haenszel chi-square test statistic; Test type: Superiority; p = 0.015, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Binimetinib (MEK162) vs Dacarbazine; Confirmed ORR + Unconfirmed ORR: The p-value (2-sided) was computed from stratified Cochran-Mantel-Haenszel chi-square test statistic; Test type: Superiority; p = 0.002, Cochran-Mantel-Haenszel

4. Secondary Outcome: Time to Response (TTR)
Description: TTR: time between date of randomization until first documented response of CR or PR. RECIST V1.1, a) CR: disappearance of all lesions; any pathological lymph nodes (TLs) or non-pathological (non-TLs) must have reduction in short axis to <10 mm; normalization of tumor marker level for non-TLs; b) PR: >=30% decrease in sum of diameter (dia) of all TLs, referring baseline sum of dia; c) PD: >=20% increase in sum of diameter of all measured TLs taking as reference smallest sum of diameter of all TLs recorded at or after baseline, sum must also be absolute increase of >=5 mm. Unequivocal progression of existing non-TLs. Appearance of >=1 new lesion. Participants who did not achieve PR or CR censored at last adequate tumor assessment date when they did not have PFS event (time from date of randomization to date of first documented PD or death due to any cause, whichever occur first) or at maximum follow-up when they had PFS event.
Time Frame: as for outcome 3
Population: Analysis population consisted of all randomized participants and who had at least once CR or PR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Binimetinib (MEK162) | Dacarbazine
Number analyzed (Participants) | 61 | 13
Months | 1.45 [1.45 to 1.48] | 2.79 [1.22 to 3.38]

5. Secondary Outcome: Duration of Objective Response (DOR)
Description: DOR: time from date of first documented response (CR or PR) to first documented progression or death due to underlying cancer. RECIST V1.1, a) CR: disappearance of all lesions; any pathological lymph nodes (TLs) or non-pathological (non-TLs) must have reduction in short axis to <10 mm; normalization of tumor marker level for non-TLs; b) PR: >=30% decrease in sum of diameter (dia) of all TLs, referring baseline sum of dia; c) PD: >=20% increase in sum of diameter of all measured target lesions taking as reference smallest sum of diameter of all target lesions recorded at or after baseline, sum must also be absolute increase of >=5 mm. Unequivocal progression of existing non-target lesions. Appearance of at least 1 new lesion. If a participant with a CR or PR had no PD or death due to underlying cancer, participants was censored at date of last adequate tumor assessment.
Time Frame: From the date of first documented response (CR or PR) to the first documented progression or death (maximum up to 77 weeks for binimetinib arm; maximum up to 61 weeks for dacarbazine arm)
Population: Analysis population consisted of all randomized participants and who had confirmed responses (CR or PR).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Binimetinib (MEK162) | Dacarbazine
Number analyzed (Participants) | 41 | 9
Months | 6.87 [4.21 to 11.07] | NA [4.14 to NA] — Median and 95% CI upper limit was not estimable due to very less number of participants with event.

6. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was calculated as the percentage of participants with a BOR of CR, PR, SD RECIST V1.1, a) CR: disappearance of all lesions; any pathological lymph nodes (TLs) or non-pathological (non-TLs) must have reduction in short axis to <10 mm; normalization of tumor marker level for non-TLs; b) PR: >=30% decrease in sum of diameter of all target lesions, taking as reference the baseline sum of diameters; c) SD: neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for PD taking as reference the smallest sum diameters; d) PD: >=20% increase in sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline, sum must also be absolute increase of >=5 mm. Unequivocal progression of existing non-target lesions. Appearance of at least 1 new lesion.
Time Frame: From date of randomization until first documented response of CR, PR, SD or non-CR/non-PD (maximum up to 77 weeks for binimetinib arm; maximum up to 61 weeks for dacarbazine arm)
Population: FAS consisted of all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Binimetinib (MEK162) | Dacarbazine
Number analyzed (Participants) | 269 | 133
Percentage of participants | 58.4 [52.2 to 64.3] | 24.8 [17.7 to 33.0]

7. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship with the study treatment. SAE was defined as one of the following: was fatal or life-threatening; resulted in persistent or significant disability/incapacity; constituted a congenital anomaly/birth defect; was medically significant; required inpatient hospitalization or prolongation of existing hospitalization. Treatment-emergent AE was defined as an AE with onset date occurring during the on-treatment period. AEs included all SAEs and non-SAEs.
Time Frame: From baseline up to 219.4 weeks for binimetinib arm; From baseline up to 123.9 weeks for dacarbazine arm
Population: The safety set consisted all participants who received at least one dose of the study drug and had at least one valid post-baseline safety evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | Binimetinib (MEK162) | Dacarbazine
Number analyzed (Participants) | 269 | 114
Participants
  AEs | 269 | 104
  SAEs | 95 | 26

8. Secondary Outcome: Number of Participants With Clinically Notable Hematology Shifts Based on National Cancer Institute Common Terminology Criteria (NCI-CTCAE) Grade, Version 4.03
Description: Clinically notable shifts are defined as worsening by at least 2 grades or to >= grade 3. Severity was graded as Grade 1: asymptomatic or mild symptoms, clinical or diagnostic observations only, intervention not indicated; Grade 2: moderate, minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental activities of daily life (ADL); Grade 3: severe or medically significant but not immediately life-threatening, hospitalization or prolongation of existing hospitalization indicated, disabling, limiting self-care ADL; Grade 4: life-threatening consequence, urgent intervention indicated; Grade 5: death related to AE.
Time Frame: From baseline up to 77 weeks in binimetinib arm; From baseline up to 61 weeks for dacarbazine arm
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Binimetinib (MEK162) | Dacarbazine
Number analyzed (Participants) | 269 | 114
Participants
  Activated partial thromboplastin time prolonged | 7 | 2
  Hemoglobin decreased | 17 | 13
  Prothrombin international normalized ratio increased | 9 | 0
  Lymphocytes increased | 20 | 0
  Lymphocytes decreased | 35 | 19
  Neutrophils decreased | 8 | 21
  Platelets decreased | 3 | 17
  Leukocytes increased | 0 | 0
  Leukocytes decreased | 6 | 26

9. Secondary Outcome: Number of Participants With Clinically Notable Clinical Chemistry/Biochemistry Shifts Based on NCI-CTCAE Grade, Version 4.03
Description: Clinically notable shifts are defined as worsening by at least 2 grades or to >= grade 3. Severity was graded as Grade 1: asymptomatic or mild symptoms, clinical or diagnostic observations only, intervention not indicated; Grade 2: moderate, minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental ADL; Grade 3: severe or medically significant but not immediately life-threatening, hospitalization or prolongation of existing hospitalization indicated, disabling, limiting self-care ADL; Grade 4: life-threatening consequence, urgent intervention indicated; Grade 5: death related to AE.
Time Frame: From baseline up to 77 weeks in binimetinib arm; From baseline up to 61 weeks for dacarbazine arm
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Binimetinib (MEK162) | Dacarbazine
Number analyzed (Participants) | 269 | 114
Participants
  Albumin decreased | 27 | 5
  Alkaline phosphatase | 8 | 2
  Alanine aminotransferase | 14 | 4
  Aspartate aminotransferase | 20 | 1
  Bilirubin | 1 | 1
  Corrected Calcium increased | 2 | 4
  Corrected Calcium decreased | 2 | 0
  Creatinine | 9 | 2
  Gamma-glutamyl transferase | 9 | 7
  Glucose serum fasting increased | 13 | 5
  Glucose serum fasting decreased | 6 | 0
  Potassium increased | 13 | 3
  Potassium decreased | 14 | 1
  Magnesium increased | 1 | 0
  Magnesium decreased | 1 | 0
  Phosphate decreased | 17 | 5
  Sodium increased | 23 | 4
  Sodium decreased | 4 | 0

10. Secondary Outcome: Number of Participants With Clinically Notable Vital Signs
Description: Abnormalities criteria included: low/high pulse rate (beats per minute [bpm]):<=50bpm with decrease from baseline >=15bpm/>=120bpm with increase from baseline >=15bpm; Low/high systolic blood pressure (millimeters of mercury [mmHg]): <=90mmHg with decrease from baseline >=20mmHg/>=160mmHg with increase from baseline >=20mmHg; Low/high diastolic blood pressure [mmHg]: <=50mmHg with decrease from baseline >=15mmHg/>=100mmHg with increase from baseline >=15mmHg; Low/high body weight (kilogram [kg]): >=20% decrease from baseline / >=10% increase from baseline; Low/high body temperature (degree Celsius [°C]): <=36°C / >= 37.5°C
Time Frame: From baseline up to 77 weeks in binimetinib arm; From baseline up to 61 weeks for dacarbazine arm
Population: The safety set consisted all participants who received at least one dose of the study drug and had at least one valid post-baseline safety evaluation. Here, "number analyzed" signifies participants evaluable for this outcome measure for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Binimetinib (MEK162) | Dacarbazine
Number analyzed (Participants) | 269 | 114
Participants
  Sitting Pulse Rate - High: number analyzed (Participants) | 260 | 106
  Sitting Pulse Rate - High | 4 | 1
  Sitting Pulse Rate - Low: number analyzed (Participants) | 259 | 105
  Sitting Pulse Rate - Low | 3 | 1
  Sitting systolic blood pressure - High: number analyzed (Participants) | 249 | 102
  Sitting systolic blood pressure - High | 43 | 8
  Sitting systolic blood pressure -Low: number analyzed (Participants) | 260 | 105
  Sitting systolic blood pressure -Low | 2 | 4
  Sitting diastolic blood pressure - High: number analyzed (Participants) | 258 | 104
  Sitting diastolic blood pressure - High | 28 | 4
  Sitting diastolic blood pressure - Low: number analyzed (Participants) | 260 | 105
  Sitting diastolic blood pressure - Low | 2 | 1
  Weight - High: number analyzed (Participants) | 261 | 105
  Weight - High | 16 | 1
  Weight - Low: number analyzed (Participants) | 261 | 105
  Weight - Low | 0 | 0
  Body temperature - High: number analyzed (Participants) | 258 | 105
  Body temperature - High | 15 | 6
  Body temperature - Low: number analyzed (Participants) | 198 | 79
  Body temperature - Low | 90 | 24

11. Secondary Outcome: Number of Participants With Notable Electrocardiogram (ECG) Values
Description: Criteria for notable ECG values were as follow: QT interval (in millisecond [msec]) new (newly occurring post-baseline value) greater than (>) 450, 480, 500, increase from baseline >30, increase from baseline >60; corrected QT interval by Fredericia formula (QTcF) in msec new (newly occurring post-baseline value) > 450, 480, 500, increase from baseline >30, increase from baseline >60; corrected QT interval by Bazett's formula (QTcB) in msec new (newly occurring post-baseline value) > 450, 480, 500, increase from baseline >30, increase from baseline >60; heart rate in bpm new (newly occurring post-baseline value) <60 and >100.
Time Frame: From baseline up to 77 weeks in binimetinib arm; From baseline up to 61 weeks for dacarbazine arm
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Binimetinib (MEK162) | Dacarbazine
Number analyzed (Participants) | 269 | 114
Participants
  QT - New > 450 msec: number analyzed (Participants) | 249 | 102
  QT - New > 450 msec | 32 | 8
  QT - New > 480 msec: number analyzed (Participants) | 259 | 103
  QT - New > 480 msec | 7 | 1
  QT - New > 500 msec: number analyzed (Participants) | 260 | 103
  QT - New > 500 msec | 5 | 0
  QT - Increase from baseline > 30 msec: number analyzed (Participants) | 261 | 103
  QT - Increase from baseline > 30 msec | 109 | 33
  QT - Increase from baseline > 60 msec: number analyzed (Participants) | 261 | 103
  QT - Increase from baseline > 60 msec | 28 | 5
  QTcF - New > 450 msec: number analyzed (Participants) | 243 | 101
  QTcF - New > 450 msec | 29 | 15
  QTcF - New > 480 msec: number analyzed (Participants) | 261 | 105
  QTcF - New > 480 msec | 10 | 1
  QTcF - New > 500 msec: number analyzed (Participants) | 262 | 106
  QTcF - New > 500 msec | 5 | 1
  QTcF - Increase from baseline > 30 msec: number analyzed (Participants) | 262 | 106
  QTcF - Increase from baseline > 30 msec | 52 | 25
  QTcF - Increase from baseline > 60 msec: number analyzed (Participants) | 262 | 106
  QTcF - Increase from baseline > 60 msec | 9 | 5
  QTcB - New > 450 msec: number analyzed (Participants) | 217 | 82
  QTcB - New > 450 msec | 65 | 26
  QTcB - New > 480 msec: number analyzed (Participants) | 250 | 100
  QTcB - New > 480 msec | 24 | 8
  QTcB - New > 500 msec: number analyzed (Participants) | 253 | 101
  QTcB - New > 500 msec | 6 | 6
  QTcB - Increase from baseline > 30 msec: number analyzed (Participants) | 255 | 102
  QTcB - Increase from baseline > 30 msec | 76 | 36
  QTcB - Increase from baseline > 60 msec: number analyzed (Participants) | 255 | 102
  QTcB - Increase from baseline > 60 msec | 11 | 9
  Heart rate - New < 60 bpm: number analyzed (Participants) | 219 | 85
  Heart rate - New < 60 bpm | 85 | 13
  Heart rate - New > 100 bpm: number analyzed (Participants) | 255 | 93
  Heart rate - New > 100 bpm | 18 | 16

12. Secondary Outcome: Number of Participants With Adverse Events of Special Interest: Cardiac Events
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship with the study treatment. Grade 1: asymptomatic or mild symptoms, clinical or diagnostic observations only, intervention not indicated; Grade 2: moderate, minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental activities of daily life (ADL); Grade 3: severe or medically significant but not immediately life-threatening, hospitalization or prolongation of existing hospitalization indicated, disabling, limiting self-care ADL; Grade 4: life-threatening consequence, urgent intervention indicated; Grade 5: death related to AE. Here, in this outcome measure data is reported for events falling in any of the grades.
Time Frame: From baseline up to 77 weeks in binimetinib arm; From baseline up to 61 weeks for dacarbazine arm
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Binimetinib (MEK162) | Dacarbazine
Number analyzed (Participants) | 269 | 114
Participants | 35 | 2

13. Secondary Outcome: Number of Participants With Clinically Significant Findings in Physical Examination
Description: A complete physical examination included the examination of general appearance, skin, neck (including thyroid), eyes, ears, nose, throat, lungs, heart, abdomen, back, lymph nodes, extremities, vascular and neurological systems. If indicated based on medical history and/or symptoms, rectal, external genitalia, breast, and pelvic examinations were performed. Clinical significance in physical examination was reported as adverse events.
Time Frame: From baseline up to 77 weeks in binimetinib arm; From baseline up to 61 weeks for dacarbazine arm
Population: No data was collected and analyzed for this outcome measure, any clinically significant physical examination findings were counted as adverse events and reported in safety section.
Arm/Group | Binimetinib (MEK162) | Dacarbazine
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Number of Participants With Adverse Events of Special Interest: Ocular Events
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship with the study treatment. Grade 1: Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated; Grade 2: Moderate; minimal, local or noninvasive intervention indicated; limiting age appropriate instrumental ADL; Grade 3: Severe or medically significant but not immediately sight threatening; Hospitalization or prolongation of existing hospitalization indicated; disabling; limiting self-care ADL; Grade 4: Sight-threatening consequences; urgent intervention indicated; blindness (20/200 or worse) in the affected eye. Here, in this outcome measure data is reported for events falling in any of the grades.
Time Frame: From baseline up to 77 weeks in binimetinib arm; From baseline up to 61 weeks for dacarbazine arm
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Binimetinib (MEK162) | Dacarbazine
Number analyzed (Participants) | 269 | 114
Participants | 6 | 0

15. Secondary Outcome: Plasma Concentration of Binimetinib
Time Frame: Day 1 of Week 1: Pre-dose, 1, 1.5, 2, 10 hours post-dose; Day 1 of Weeks 4, 7: Pre-dose, 1.5 hours post-dose; Day 1 of Weeks 10, 13: Pre-dose
Population: The pharmacokinetic analysis set (PAS) consisted of all participants who received at least one dose of binimetinib and had at least one evaluable post-baseline binimetinib concentration measurement. Here, "Overall Number of Participants Analyzed" = number of participants evaluable for this outcome measure. This outcome was planned to be evaluated only for binimetinib arm. Here, "number analyzed" signifies participants evaluable for this outcome measure for specified timeframes.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter
Arm/Group | Binimetinib (MEK162)
Number analyzed (Participants) | 264
Nanogram per milliliter
  Week 1 Day 1, Pre-dose: number analyzed (Participants) | 253
  Week 1 Day 1, Pre-dose | 64.4 (1132.3)
  Week 1 Day 1, 1 hour (hr) Post-dose: number analyzed (Participants) | 223
  Week 1 Day 1, 1 hour (hr) Post-dose | 182 (237.6)
  Week 1 Day 1, 1.5 hr Post-dose: number analyzed (Participants) | 217
  Week 1 Day 1, 1.5 hr Post-dose | 313 (71.6)
  Week 1 Day 1, 2 hr Post-dose: number analyzed (Participants) | 26
  Week 1 Day 1, 2 hr Post-dose | 321 (64.4)
  Week 1 Day 1, 10 hr Post-dose: number analyzed (Participants) | 245
  Week 1 Day 1, 10 hr Post-dose | 153 (52.6)
  Week 4 Day 1, Pre-dose: number analyzed (Participants) | 161
  Week 4 Day 1, Pre-dose | 101 (100.8)
  Week 4 Day 1, 1.5 hr Post-dose: number analyzed (Participants) | 155
  Week 4 Day 1, 1.5 hr Post-dose | 418 (51.9)
  Week 7 Day 1, Pre-dose: number analyzed (Participants) | 133
  Week 7 Day 1, Pre-dose | 101 (97.7)
  Week 7 Day 1, 1.5 hr Post-dose: number analyzed (Participants) | 134
  Week 7 Day 1, 1.5 hr Post-dose | 372 (63.4)
  Week 10 Day 1, Pre-dose: number analyzed (Participants) | 80
  Week 10 Day 1, Pre-dose | 92.9 (60.6)
  Week 13 Day 1, Pre-dose: number analyzed (Participants) | 53
  Week 13 Day 1, Pre-dose | 93.9 (89.8)

16. Secondary Outcome: Time to Definitive 10% Deterioration in Global Health Status Score of European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 (QLQ-C30)
Description: The time to definitive 10% deterioration was defined as the time from the date of randomization to the date of event, which was defined as death due to any cause or at least 10% worsening of the corresponding scale score, relative to baseline, with no later improvement above this threshold observed during the course of the study or death due to any cause. If a participant had no event prior to analysis cut-off or start of another anticancer therapy, time to deterioration was censored at the date of the last adequate health related quality of life (HRQoL) evaluation. EORTC QLQ-C30: 5 functional scales (physical, role, cognitive, emotional, and social), a global health status scale, 3 symptom scales (nausea/vomiting, pain, fatigue) and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea and financial difficulties). All scales and single-item measures range =0 to 100. High score for global health status = high quality of life.
Time Frame: From baseline up to 77 weeks in binimetinib arm; From baseline up to 61 weeks for dacarbazine arm
Population: FAS consisted of all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Binimetinib (MEK162) | Dacarbazine
Number analyzed (Participants) | 269 | 133
Months | 2.79 [1.64 to 4.24] | 4.27 [2.86 to NA] — 95% CI upper limit was not estimable due to very less number of participants with event.
Statistical Analysis 1: Comparison: Binimetinib (MEK162) vs Dacarbazine; Test type: Superiority; Log Rank; Hazard Ratio (HR) = 1.43, 95% CI 2-sided [0.96 to 2.13]

17. Secondary Outcome: Change From Baseline in Global Health Status Score of EORTC QLQ-C30 at Weeks 4, 7, 13, 19, 25, 34, 43, 52, 61, 70, End of Treatment, Safety Follow-up Visit, Post-Treatment Follow-up Visit 1, 2, 3, 4, 5 and 6
Description: EORTC QLQ-C30: 5 functional scales (physical, role, cognitive, emotional, and social), a h global health status scale, 3 symptom scales (nausea/vomiting, pain, fatigue) and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea and financial difficulties). All scales and single-item measures range =0 to 100. High score for global health status = high quality of life. Post-treatment tumor assessments follow up visits occurred at every 9 weeks if participants started new anticancer therapy.
Time Frame: Both arms: Baseline, Day 1 Treatment Week (TW) 4,7,13,19,25,34,43,52; Post-treatment follow-up Visit (FUV) 1 to 6; Binimetinib: Day 1 TW61,70; End of treatment (EOT= TW73); Safety FUV=30 days post TW73; Dacarbazine: EOT=TW 57;Safety FUV=30 days post TW57
Population: FAS consisted of all randomized participants. Here, "Number analyzed" signifies number of participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Binimetinib (MEK162) | Dacarbazine
Number analyzed (Participants) | 269 | 133
Units on a scale
  Baseline: number analyzed (Participants) | 257 | 113
  Baseline | 68.35 (23.463) | 70.50 (21.823)
  Week 4 Day 1: number analyzed (Participants) | 223 | 83
  Week 4 Day 1 | -5.75 (22.285) | -1.81 (17.512)
  Week 7 Day 1: number analyzed (Participants) | 200 | 67
  Week 7 Day 1 | -8.63 (22.562) | 0.00 (15.691)
  Week 13 Day 1: number analyzed (Participants) | 146 | 31
  Week 13 Day 1 | -8.28 (19.659) | -1.34 (16.955)
  Week 19 Day 1: number analyzed (Participants) | 87 | 23
  Week 19 Day 1 | -8.05 (21.053) | -3.26 (22.296)
  Week 25 Day 1: number analyzed (Participants) | 52 | 12
  Week 25 Day 1 | -10.58 (21.775) | -3.47 (13.036)
  Week 34 Day 1: number analyzed (Participants) | 24 | 7
  Week 34 Day 1 | -6.25 (18.755) | 3.57 (20.893)
  Week 43 Day 1: number analyzed (Participants) | 11 | 6
  Week 43 Day 1 | -11.36 (20.841) | -6.94 (23.224)
  Week 52 Day 1: number analyzed (Participants) | 11 | 2
  Week 52 Day 1 | -1.52 (20.006) | -8.33 (11.785)
  Week 61 Day 1: number analyzed (Participants) | 5 | 0
  Week 61 Day 1 | -10.00 (18.066) |
  Week 70 Day 1: number analyzed (Participants) | 2 | 0
  Week 70 Day 1 | -20.83 (5.893) |
  End of Treatment: number analyzed (Participants) | 209 | 89
  End of Treatment | -12.20 (22.512) | -6.74 (21.536)
  30-day safety follow-up: number analyzed (Participants) | 71 | 13
  30-day safety follow-up | -8.10 (21.361) | -9.62 (14.372)
  Post treatment follow-up 1: number analyzed (Participants) | 21 | 32
  Post treatment follow-up 1 | -5.95 (19.211) | -8.59 (21.218)
  Post treatment follow-up 2: number analyzed (Participants) | 1 | 0
  Post treatment follow-up 2 | 0.00 (NA) — SD was not estimable due to very less number of participants with event. |
  Post treatment follow-up 3: number analyzed (Participants) | 1 | 0
  Post treatment follow-up 3 | 16.67 (NA) — SD was not estimable due to very less number of participants with event. |
  Post treatment follow-up 4: number analyzed (Participants) | 2 | 0
  Post treatment follow-up 4 | 25.00 (11.785) |
  Post treatment follow-up 5: number analyzed (Participants) | 2 | 0
  Post treatment follow-up 5 | 25.00 (11.785) |
  Post treatment follow-up 6: number analyzed (Participants) | 1 | 0
  Post treatment follow-up 6 | 33.33 (NA) — SD was not estimable due to very less number of participants with event. |

18. Secondary Outcome: Change From Baseline in EuroQoL-5 Dimensions- 5 Levels (EQ-5D-5L) Index Score at Weeks 4, 7, 13, 19, 25, 34, 43, 52, 61, 70, End of Treatment, Safety Follow-up Visit, Post-treatment Follow-up Visit 1, 2, 3, 4, 5 and 6
Description: EQ-5D-5L, is a standardized measure of health utility that provides a single index value for one's health status. EQ-5D-5L contained 1 item for each of 5 dimensions: mobility, self-care, usual activities, pain/discomfort, anxiety/depression. Each dimension has 5 levels: 1= no problems, 2= slight problems, 3= moderate problems, 4= severe problems, and 5= extreme problems. Index score: participant responses to the 5 dimensions reflected a specific health state that corresponded to a population preference weight for that state on a continuous scale of 0 (death) to 1 (perfect health). Higher index scores = better health state. Post-treatment tumor assessments follow up visits occurred at every 9 weeks if participants started new anticancer therapy.
Time Frame: as for outcome 17
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Binimetinib (MEK162) | Dacarbazine
Number analyzed (Participants) | 269 | 133
Units on a scale
  Baseline: number analyzed (Participants) | 257 | 112
  Baseline | 0.7780 (0.22464) | 0.7657 (0.23003)
  Week 4 Day 1: number analyzed (Participants) | 221 | 83
  Week 4 Day 1 | -0.0422 (0.18291) | 0.0110 (0.12135)
  Week 7 Day 1: number analyzed (Participants) | 201 | 67
  Week 7 Day 1 | -0.0397 (0.19154) | 0.0132 (0.14084)
  Week 13 Day 1: number analyzed (Participants) | 145 | 32
  Week 13 Day 1 | -0.0773 (0.17543) | 0.0198 (0.15236)
  Week 19 Day 1: number analyzed (Participants) | 90 | 23
  Week 19 Day 1 | -0.0576 (0.22503) | 0.0257 (0.18052)
  Week 25 Day 1: number analyzed (Participants) | 55 | 12
  Week 25 Day 1 | -0.1563 (0.32142) | 0.0657 (0.16052)
  Week 34 Day 1: number analyzed (Participants) | 25 | 6
  Week 34 Day 1 | -0.0801 (0.11141) | 0.0617 (0.15254)
  Week 43 Day 1: number analyzed (Participants) | 12 | 6
  Week 43 Day 1 | -0.0170 (0.22978) | 0.1060 (0.15033)
  Week 52 Day 1: number analyzed (Participants) | 11 | 2
  Week 52 Day 1 | -0.0389 (0.24609) | 0.0000 (0.00000)
  Week 61 Day 1: number analyzed (Participants) | 5 | 0
  Week 61 Day 1 | 0.0690 (0.21080) |
  Week 70 Day 1: number analyzed (Participants) | 2 | 0
  Week 70 Day 1 | 0.0120 (0.14001) |
  End of Treatment: number analyzed (Participants) | 210 | 90
  End of Treatment | -0.0978 (0.23931) | -0.0540 (0.19164)
  30-day safety follow-up: number analyzed (Participants) | 71 | 13
  30-day safety follow-up | -0.1165 (0.24410) | -0.0740 (0.17682)
  Post treatment follow-up 1: number analyzed (Participants) | 22 | 32
  Post treatment follow-up 1 | -0.0820 (0.11993) | -0.0438 (0.25374)
  Post treatment follow-up 2: number analyzed (Participants) | 1 | 0
  Post treatment follow-up 2 | -0.2480 (NA) — SD was not estimable due to very less number of participants with event. |
  Post treatment follow-up 3: number analyzed (Participants) | 1 | 0
  Post treatment follow-up 3 | -0.1210 (NA) — SD was not estimable due to very less number of participants with event. |
  Post treatment follow-up 4: number analyzed (Participants) | 2 | 0
  Post treatment follow-up 4 | 0.1115 (0.15768) |
  Post treatment follow-up 5: number analyzed (Participants) | 2 | 0
  Post treatment follow-up 5 | 0.1730 (0.24466) |
  Post treatment follow-up 6: number analyzed (Participants) | 1 | 0
  Post treatment follow-up 6 | 0.2230 (NA) — SD was not estimable due to very less number of participants with event. |

19. Secondary Outcome: Time to Definitive 1 Point Deterioration in Eastern Cooperative Oncology Group (ECOG) Performance Status (PS)
Description: ECOG PS was used to assess the physical health of participants, and ranged from 0 (most active) to 5 (dead). ECOG PS grades: 0= fully active, able to carry on all pre-disease performance without restriction, 1= restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work, 2= ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours, 3= capable of only limited self-care, confined to bed or chair more than 50% of waking hours, 4=completely disabled. cannot carry on any selfcare. Totally confined to bed or chair and 5= dead. Definitive deterioration is defined as on treatment death due to any cause or decrease in ECOG PS by at least one category from baseline score.
Time Frame: From baseline up to 73 weeks 3 days for binimetinib arm; From baseline up to 57 weeks 3 days for dacarbazine arm
Population: The safety set consisted all participants who received at least one dose of the study drug and had at least one valid post-baseline safety evaluation. Here, "Overall Number of Participants Analyzed" = number of participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Binimetinib (MEK162) | Dacarbazine
Number analyzed (Participants) | 262 | 105
Months | NA [5.62 to NA] — Median and upper limit of 95% CI, was not estimable due to very less number of participants with event. | NA [NA to NA] — Data was not estimable due to very less number of participants with event.
Statistical Analysis 1: Comparison: Binimetinib (MEK162) vs Dacarbazine; Log-rank test and Cox PH model were stratified by American joint committee on cancer stage, prior line immunotherapy and ECOG performance status. P-value was one tailed and was based on the log-rank score test. Hazard ratio and 95% CI was based on a Wald test from Cox model; Test type: Superiority; p = 0.995, Log Rank; Hazard Ratio (HR) = 2.20, 95% CI 2-sided [1.19 to 4.06]

20. Secondary Outcome: Number of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Status (PS)
Description: ECOG PS was used to assess the physical health of participants, and ranged from 0 (most active) to 5 (dead). ECOG PS grades: 0= fully active, able to carry on all pre-disease performance without restriction, 1= restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work, 2= ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours, 3= capable of only limited self-care, 4=completely disabled. cannot carry on any selfcare. Totally confined to bed or chair confined to bed or chair more than 50% of waking hours and 5= dead. Post-treatment tumor assessments follow up visits occurred at every 9 weeks if participants started new anticancer therapy.
Time Frame: For both arms: Baseline, Weeks 4, 7, 10, 13, 16, 19, 22, 25, 28, 31, 34, 37, 40, 43, 46, 49, 52, 55 and 30-day Follow-up For binimetinib only: Weeks 58, 61, 64, 67, 70, 73
Population: The safety set consisted all participants who received at least one dose of the study drug and had at least one valid post-baseline safety evaluation. Here, "Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Binimetinib (MEK162) | Dacarbazine
Number analyzed (Participants) | 269 | 114
Participants
  Baseline : Grade 0 | 193 | 82
  Baseline: Grade 1 | 76 | 31
  Baseline : Grade 2 | 0 | 1
  Week 4 Day 1: Grade 0: number analyzed (Participants) | 256 | 97
  Week 4 Day 1: Grade 0 | 146 | 66
  Week 4 Day 1: Grade 1: number analyzed (Participants) | 256 | 97
  Week 4 Day 1: Grade 1 | 101 | 27
  Week 4 Day 1: Grade 2: number analyzed (Participants) | 256 | 97
  Week 4 Day 1: Grade 2 | 6 | 4
  Week 4 Day 1: Grade 3: number analyzed (Participants) | 256 | 97
  Week 4 Day 1: Grade 3 | 3 | 0
  Week 7 Day 1: Grade 0: number analyzed (Participants) | 236 | 80
  Week 7 Day 1: Grade 0 | 138 | 51
  Week 7 Day 1: Grade 1: number analyzed (Participants) | 236 | 80
  Week 7 Day 1: Grade 1 | 84 | 26
  Week 7 Day 1: Grade 2: number analyzed (Participants) | 236 | 80
  Week 7 Day 1: Grade 2 | 10 | 3
  Week 7 Day 1: Grade 3: number analyzed (Participants) | 236 | 80
  Week 7 Day 1: Grade 3 | 3 | 0
  Week 7 Day 1: Grade 4: number analyzed (Participants) | 236 | 80
  Week 7 Day 1: Grade 4 | 1 | 0
  Week 10 Day 1: Grade 0: number analyzed (Participants) | 201 | 51
  Week 10 Day 1: Grade 0 | 118 | 34
  Week 10 Day 1: Grade 1: number analyzed (Participants) | 201 | 51
  Week 10 Day 1: Grade 1 | 72 | 15
  Week 10 Day 1: Grade 2: number analyzed (Participants) | 201 | 51
  Week 10 Day 1: Grade 2 | 8 | 2
  Week 10 Day 1: Grade 3: number analyzed (Participants) | 201 | 51
  Week 10 Day 1: Grade 3 | 3 | 0
  Week 13 Day 1: Grade 0: number analyzed (Participants) | 167 | 43
  Week 13 Day 1: Grade 0 | 93 | 29
  Week 13 Day 1: Grade 1: number analyzed (Participants) | 167 | 43
  Week 13 Day 1: Grade 1 | 62 | 14
  Week 13 Day 1: Grade 2: number analyzed (Participants) | 167 | 43
  Week 13 Day 1: Grade 2 | 11 | 0
  Week 13 Day 1: Grade 3: number analyzed (Participants) | 167 | 43
  Week 13 Day 1: Grade 3 | 1 | 0
  Week 16 Day 1: Grade 0: number analyzed (Participants) | 124 | 30
  Week 16 Day 1: Grade 0 | 70 | 24
  Week 16 Day 1: Grade 1: number analyzed (Participants) | 124 | 30
  Week 16 Day 1: Grade 1 | 48 | 5
  Week 16 Day 1: Grade 2: number analyzed (Participants) | 124 | 30
  Week 16 Day 1: Grade 2 | 5 | 1
  Week 16 Day 1: Grade 4: number analyzed (Participants) | 124 | 30
  Week 16 Day 1: Grade 4 | 1 | 0
  Week 19 Day 1: Grade 0: number analyzed (Participants) | 100 | 28
  Week 19 Day 1: Grade 0 | 53 | 19
  Week 19 Day 1: Grade 1: number analyzed (Participants) | 100 | 28
  Week 19 Day 1: Grade 1 | 43 | 7
  Week 19 Day 1:Grade 2: number analyzed (Participants) | 100 | 28
  Week 19 Day 1:Grade 2 | 4 | 2
  Week 22 Day 1: Grade 0: number analyzed (Participants) | 72 | 22
  Week 22 Day 1: Grade 0 | 42 | 17
  Week 22 Day 1: Grade 1: number analyzed (Participants) | 72 | 22
  Week 22 Day 1: Grade 1 | 26 | 5
  Week 22 Day 1: Grade 2: number analyzed (Participants) | 72 | 22
  Week 22 Day 1: Grade 2 | 3 | 0
  Week 22 Day 1: Grade 3: number analyzed (Participants) | 72 | 22
  Week 22 Day 1: Grade 3 | 1 | 0
  Week 25 Day 1: Grade 0: number analyzed (Participants) | 58 | 19
  Week 25 Day 1: Grade 0 | 37 | 13
  Week 25 Day 1: Grade 1: number analyzed (Participants) | 58 | 19
  Week 25 Day 1: Grade 1 | 19 | 6
  Week 25 Day 1: Grade 2: number analyzed (Participants) | 58 | 19
  Week 25 Day 1: Grade 2 | 1 | 0
  Week 25 Day 1: Grade 3: number analyzed (Participants) | 58 | 19
  Week 25 Day 1: Grade 3 | 1 | 0
  Week 28 Day 1: Grade 0: number analyzed (Participants) | 46 | 11
  Week 28 Day 1: Grade 0 | 28 | 9
  Week 28 Day 1: Grade 1: number analyzed (Participants) | 46 | 11
  Week 28 Day 1: Grade 1 | 15 | 2
  Week 28 Day 1: Grade 2: number analyzed (Participants) | 46 | 11
  Week 28 Day 1: Grade 2 | 2 | 0
  Week 28 Day 1: Grade 5: number analyzed (Participants) | 46 | 11
  Week 28 Day 1: Grade 5 | 1 | 0
  Week 31 Day 1: Grade 0: number analyzed (Participants) | 34 | 9
  Week 31 Day 1: Grade 0 | 22 | 7
  Week 31 Day 1: Grade 1: number analyzed (Participants) | 34 | 9
  Week 31 Day 1: Grade 1 | 11 | 2
  Week 31 Day 1: Grade 2: number analyzed (Participants) | 34 | 9
  Week 31 Day 1: Grade 2 | 1 | 0
  Week 34 Day 1: Grade 0: number analyzed (Participants) | 29 | 10
  Week 34 Day 1: Grade 0 | 20 | 9
  Week 34 Day 1: Grade 1: number analyzed (Participants) | 29 | 10
  Week 34 Day 1: Grade 1 | 7 | 1
  Week 34 Day 1: Grade 2: number analyzed (Participants) | 29 | 10
  Week 34 Day 1: Grade 2 | 2 | 0
  Week 37 Day 1: Grade 0: number analyzed (Participants) | 20 | 8
  Week 37 Day 1: Grade 0 | 16 | 7
  Week 37 Day 1: Grade 1: number analyzed (Participants) | 20 | 8
  Week 37 Day 1: Grade 1 | 4 | 1
  Week 40 Day 1: Grade 0: number analyzed (Participants) | 15 | 7
  Week 40 Day 1: Grade 0 | 15 | 6
  Week 40 Day 1: Grade 1: number analyzed (Participants) | 15 | 7
  Week 40 Day 1: Grade 1 | 0 | 1
  Week 43 Day 1: Grade 0: number analyzed (Participants) | 14 | 5
  Week 43 Day 1: Grade 0 | 12 | 5
  Week 43 Day 1: Grade 1: number analyzed (Participants) | 14 | 5
  Week 43 Day 1: Grade 1 | 1 | 0
  Week 43 Day 1: Grade 2: number analyzed (Participants) | 14 | 5
  Week 43 Day 1: Grade 2 | 1 | 0
  Week 46 Day 1: Grade 0: number analyzed (Participants) | 14 | 4
  Week 46 Day 1: Grade 0 | 11 | 4
  Week 46 Day 1: Grade 1: number analyzed (Participants) | 14 | 4
  Week 46 Day 1: Grade 1 | 2 | 0
  Week 46 Day 1: Grade 2: number analyzed (Participants) | 14 | 4
  Week 46 Day 1: Grade 2 | 1 | 0
  Week 49 Day 1: Grade 0: number analyzed (Participants) | 11 | 1
  Week 49 Day 1: Grade 0 | 9 | 1
  Week 49 Day 1: Grade 1: number analyzed (Participants) | 11 | 1
  Week 49 Day 1: Grade 1 | 2 | 0
  Week 52 Day 1: Grade 0: number analyzed (Participants) | 11 | 3
  Week 52 Day 1: Grade 0 | 10 | 2
  Week 52 Day 1: Grade 1: number analyzed (Participants) | 11 | 3
  Week 52 Day 1: Grade 1 | 1 | 1
  Week 55 Day 1: Grade 0: number analyzed (Participants) | 10 | 2
  Week 55 Day 1: Grade 0 | 9 | 1
  Week 55 Day 1: Grade 1: number analyzed (Participants) | 10 | 2
  Week 55 Day 1: Grade 1 | 1 | 1
  Week 58 Day 1: Grade 0: number analyzed (Participants) | 8 | 0
  Week 58 Day 1: Grade 0 | 7 |
  Week 58 Day 1: Grade 1: number analyzed (Participants) | 8 | 0
  Week 58 Day 1: Grade 1 | 1 |
  Week 61 Day 1: Grade 0: number analyzed (Participants) | 5 | 0
  Week 61 Day 1: Grade 0 | 5 |
  Week 64 Day 1: Grade 0: number analyzed (Participants) | 4 | 0
  Week 64 Day 1: Grade 0 | 4 |
  Week 67 Day 1: Grade 0: number analyzed (Participants) | 3 | 0
  Week 67 Day 1: Grade 0 | 3 |
  Week 70 Day 1: Grade 0: number analyzed (Participants) | 2 | 0
  Week 70 Day 1: Grade 0 | 2 |
  Week 73 Day 1: Grade 0: number analyzed (Participants) | 1 | 0
  Week 73 Day 1: Grade 0 | 1 |
  Safety Follow up Visit: Grade 0: number analyzed (Participants) | 105 | 44
  Safety Follow up Visit: Grade 0 | 42 | 24
  Safety Follow up Visit: Grade 1: number analyzed (Participants) | 105 | 44
  Safety Follow up Visit: Grade 1 | 41 | 16
  Safety Follow up Visit: Grade 2: number analyzed (Participants) | 105 | 44
  Safety Follow up Visit: Grade 2 | 14 | 4
  Safety Follow up Visit: Grade 3: number analyzed (Participants) | 105 | 44
  Safety Follow up Visit: Grade 3 | 4 | 0
  Safety Follow up Visit: Grade 4: number analyzed (Participants) | 105 | 44
  Safety Follow up Visit: Grade 4 | 4 | 0

21. Secondary Outcome: Number of Participants With Neuroblastoma RAS Viral (V-ras) Oncogene Homolog (NRAS) Mutation Status at Baseline
Description: Number of participants with NRAS mutation status at baseline were reported.
Time Frame: Baseline
Population: FAS consisted of all randomized participants. Here, "number analyzed" signifies participants evaluable for this outcome measure for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Binimetinib (MEK162) | Dacarbazine
Number analyzed (Participants) | 269 | 133
Participants
  Wild Type | 0 | 1
  Mutant: Q61K: number analyzed (Participants) | 269 | 132
  Mutant: Q61K | 100 | 51
  Mutant: Q61L: number analyzed (Participants) | 269 | 132
  Mutant: Q61L | 32 | 17
  Mutant: Q61R: number analyzed (Participants) | 269 | 132
  Mutant: Q61R | 137 | 64

ADVERSE EVENTS:
Time Frame: From baseline up to 219.4 weeks for binimetinib arm; From baseline up to 123.9 weeks for dacarbazine arm
Description: Same event may appear as AE and serious AE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study. Safety analysis set population included all participants who have received at least one dose of the study drug and had at least one valid post-baseline safety assessment.
Arm/Group | Binimetinib (MEK162) | Dacarbazine
Serious Adverse Events (participants affected / at risk) | 95/269 | 26/114
Other Adverse Events (participants affected / at risk) | 266/269 | 100/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Binimetinib (MEK162) (N=269) | Dacarbazine (N=114)
TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 2 | 0
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 | 1
ANAEMIA (Blood and lymphatic system disorders) | 2 | 0
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 1
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 1
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 | 2
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 0
TACHYARRHYTHMIA (Cardiac disorders) | 1 | 1
RETINAL VEIN OCCLUSION (Eye disorders) | 4 | 0
RETINAL DETACHMENT (Eye disorders) | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 2 | 0
VOMITING (Gastrointestinal disorders) | 3 | 0
MOUTH ULCERATION (Gastrointestinal disorders) | 1 | 0
MALAISE (General disorders) | 0 | 1
PYREXIA (General disorders) | 1 | 3
HEPATIC FAILURE (Hepatobiliary disorders) | 1 | 0
SEPTIC SHOCK (Infections and infestations) | 1 | 0
SKIN INFECTION (Infections and infestations) | 3 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1
MUSCLE INJURY (Injury, poisoning and procedural complications) | 1 | 0
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 3 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0
EJECTION FRACTION DECREASED (Investigations) | 1 | 0
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 1 | 0
HAEMOGLOBIN DECREASED (Investigations) | 1 | 0
INTRAOCULAR PRESSURE INCREASED (Investigations) | 1 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 2 | 0
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
MYASTHENIC SYNDROME (Nervous system disorders) | 1 | 0
PERIPHERAL SENSORIMOTOR NEUROPATHY (Nervous system disorders) | 1 | 0
LETHARGY (Nervous system disorders) | 0 | 1
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 | 0
RENAL FAILURE (Renal and urinary disorders) | 2 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 4 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 | 2
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 1 | 0
PSORIASIS (Skin and subcutaneous tissue disorders) | 1 | 0
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 | 0
HYPERTENSIVE CRISIS (Vascular disorders) | 2 | 0
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
MALIGNANT ASCITES (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 1
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 0
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 0 | 1
ANGINA PECTORIS (Cardiac disorders) | 1 | 0
ATRIAL FLUTTER (Cardiac disorders) | 1 | 0
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 1 | 0
ATRIOVENTRICULAR BLOCK FIRST DEGREE (Cardiac disorders) | 1 | 0
MITRAL VALVE DISEASE (Cardiac disorders) | 1 | 0
RETINAL VEIN THROMBOSIS (Eye disorders) | 2 | 0
CONSTIPATION (Gastrointestinal disorders) | 2 | 0
NAUSEA (Gastrointestinal disorders) | 2 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 1
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 0
ASCITES (Gastrointestinal disorders) | 1 | 0
AUTOIMMUNE PANCREATITIS (Gastrointestinal disorders) | 1 | 0
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 1 | 0
DUODENAL PERFORATION (Gastrointestinal disorders) | 1 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 1 | 0
INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 | 0
INTUSSUSCEPTION (Gastrointestinal disorders) | 1 | 0
LARGE INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0
MESENTERIC VEIN THROMBOSIS (Gastrointestinal disorders) | 1 | 0
SUBILEUS (Gastrointestinal disorders) | 1 | 0
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 10 | 0
AXILLARY PAIN (General disorders) | 1 | 0
FATIGUE (General disorders) | 1 | 0
MULTIPLE ORGAN DYSFUNCTION SYNDROME (General disorders) | 1 | 0
OEDEMA PERIPHERAL (General disorders) | 1 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 0
CHOLESTASIS (Hepatobiliary disorders) | 0 | 1
CELLULITIS (Infections and infestations) | 2 | 0
ERYSIPELAS (Infections and infestations) | 2 | 0
PYELONEPHRITIS ACUTE (Infections and infestations) | 2 | 0
SEPSIS (Infections and infestations) | 2 | 2
SOFT TISSUE INFECTION (Infections and infestations) | 2 | 0
UROSEPSIS (Infections and infestations) | 2 | 0
ABSCESS LIMB (Infections and infestations) | 1 | 0
DERMO-HYPODERMITIS (Infections and infestations) | 1 | 0
HERPES ZOSTER (Infections and infestations) | 1 | 0
OSTEOMYELITIS (Infections and infestations) | 1 | 0
PNEUMOCOCCAL SEPSIS (Infections and infestations) | 1 | 0
PNEUMONIA (Infections and infestations) | 1 | 1
VIRAL INFECTION (Infections and infestations) | 1 | 0
LUNG INFECTION (Infections and infestations) | 0 | 1
PERINEAL ABSCESS (Infections and infestations) | 0 | 1
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 1 | 0
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
BLOOD PRESSURE INCREASED (Investigations) | 1 | 0
EASTERN COOPERATIVE ONCOLOGY GROUP PERFORMANCE STATUS WORSENED (Investigations) | 1 | 0
GENERAL PHYSICAL CONDITION ABNORMAL (Investigations) | 1 | 0
DIABETIC METABOLIC DECOMPENSATION (Metabolism and nutrition disorders) | 1 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 2 | 0
INTERVERTEBRAL DISC COMPRESSION (Musculoskeletal and connective tissue disorders) | 1 | 0
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 2
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 1
SPINAL CORD COMPRESSION (Nervous system disorders) | 2 | 0
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 | 0
DROPPED HEAD SYNDROME (Nervous system disorders) | 1 | 0
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 1 | 0
MOTOR DYSFUNCTION (Nervous system disorders) | 1 | 0
SCIATICA (Nervous system disorders) | 1 | 0
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 1 | 1
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 | 0
BRAIN OEDEMA (Nervous system disorders) | 0 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 1
DEMENTIA (Nervous system disorders) | 0 | 1
ENCEPHALOPATHY (Nervous system disorders) | 0 | 1
PROGRESSIVE SUPRANUCLEAR PALSY (Nervous system disorders) | 0 | 1
NEPHROLITHIASIS (Renal and urinary disorders) | 1 | 0
HAEMORRHAGE (Vascular disorders) | 2 | 0
AORTIC DILATATION (Vascular disorders) | 1 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 | 0
EMBOLISM (Vascular disorders) | 1 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 2 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 2 | 0
ABNORMAL BEHAVIOUR (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Binimetinib (MEK162) (N=269) | Dacarbazine (N=114)
ANAEMIA (Blood and lymphatic system disorders) | 19 | 11
LYMPHOPENIA (Blood and lymphatic system disorders) | 7 | 7
NEUTROPENIA (Blood and lymphatic system disorders) | 4 | 21
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 | 17
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 8
RETINAL DETACHMENT (Eye disorders) | 35 | 0
EYELID OEDEMA (Eye disorders) | 28 | 0
VISION BLURRED (Eye disorders) | 20 | 1
SUBRETINAL FLUID (Eye disorders) | 19 | 0
MACULAR OEDEMA (Eye disorders) | 17 | 0
PERIORBITAL OEDEMA (Eye disorders) | 14 | 0
DIARRHOEA (Gastrointestinal disorders) | 109 | 15
NAUSEA (Gastrointestinal disorders) | 85 | 35
VOMITING (Gastrointestinal disorders) | 58 | 15
CONSTIPATION (Gastrointestinal disorders) | 39 | 22
ABDOMINAL PAIN (Gastrointestinal disorders) | 24 | 8
DRY MOUTH (Gastrointestinal disorders) | 22 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 16 | 3
OEDEMA PERIPHERAL (General disorders) | 97 | 5
FATIGUE (General disorders) | 68 | 38
ASTHENIA (General disorders) | 44 | 19
PYREXIA (General disorders) | 34 | 16
PERIPHERAL SWELLING (General disorders) | 15 | 2
FACE OEDEMA (General disorders) | 14 | 0
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 119 | 3
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 39 | 5
EJECTION FRACTION DECREASED (Investigations) | 35 | 2
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 23 | 8
INTRAOCULAR PRESSURE INCREASED (Investigations) | 19 | 0
WEIGHT DECREASED (Investigations) | 13 | 6
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 8 | 7
PLATELET COUNT DECREASED (Investigations) | 2 | 11
NEUTROPHIL COUNT DECREASED (Investigations) | 1 | 8
DECREASED APPETITE (Metabolism and nutrition disorders) | 34 | 19
MYALGIA (Musculoskeletal and connective tissue disorders) | 28 | 3
BACK PAIN (Musculoskeletal and connective tissue disorders) | 19 | 6
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 18 | 3
NECK PAIN (Musculoskeletal and connective tissue disorders) | 17 | 2
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 16 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 11 | 6
DYSGEUSIA (Nervous system disorders) | 21 | 2
HEADACHE (Nervous system disorders) | 18 | 9
DIZZINESS (Nervous system disorders) | 17 | 3
INSOMNIA (Psychiatric disorders) | 17 | 8
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 27 | 5
COUGH (Respiratory, thoracic and mediastinal disorders) | 20 | 10
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 106 | 1
RASH (Skin and subcutaneous tissue disorders) | 96 | 2
DRY SKIN (Skin and subcutaneous tissue disorders) | 37 | 2
PRURITUS (Skin and subcutaneous tissue disorders) | 27 | 2
SKIN FISSURES (Skin and subcutaneous tissue disorders) | 26 | 0
ALOPECIA (Skin and subcutaneous tissue disorders) | 24 | 3
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 23 | 0
ERYTHEMA (Skin and subcutaneous tissue disorders) | 17 | 2
HYPERTENSION (Vascular disorders) | 36 | 4
RASH PUSTULAR (Infections and infestations) | 18 | 0
NASOPHARYNGITIS (Infections and infestations) | 17 | 5
ERYSIPELAS (Infections and infestations) | 15 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.